CLINICAL TRIAL: NCT00893048
Title: Utility of Prednisone in the Treatment of Cellulitis
Brief Title: The Use of Oral Steroids in the Treatment of Cellulitis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study never enrolled any subjects before auto-terminated by the internal IRB.
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8876
Record Dates: First submitted 2009-05-01; First posted 2009-05-05 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Cellulitis; Erysipelas
Keywords: prednisone; cellulitis; erysipelas; steroids; oral
MeSH Terms: conditions — Cellulitis; Erysipelas | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prednisone (Experimental): Use of prednisone to decrease LOS and overall treatment time of cellulitis
  Interventions: Drug: Prednisone
- Placebo (Experimental)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Prednisone — Prednisone, 60 mg, one time at time of diagnosis
  Other Names: sterapred; sterapred DS
  Arms: Prednisone
Drug: Placebo Oral Tablet — Placebo
  Arms: Placebo

SUMMARY:
The prevalence of cellulitis in society is very high, as much as 3% of visits to Emergency Departments are for the treatment of this disease. The treatment of cellulitis varies depending on the severity. Low severity cases are treated with pain control and antibiotics by mouth and high severity are treated with antibiotics intravenously and pain control. The investigator's hypothesis is to see if the addition of steroids, which are known to decrease inflammation, will decrease the length of the disease process. If so, it will decrease the length of stay if IV antibiotics are needed, it will decrease duration of days out of work and decrease the overall pain control required and therefore patient satisfaction.

DETAILED DESCRIPTION:
The incidence of cellulitis is about 24.6 cases per 1000 person-years, which is an estimate, since cellulitis is not a reportable disease. In some Emergency Departments up to 3% of visits are for cellulitis. Depending on the severity of the disease, some are treated as outpatients, and others are admitted for IV antibiotics. In some Emergency Departments cases of cellulitis are treated in an observation area for 23 hours with doses of IV antibiotics. My proposed research is to see if the addition of one dose of prednisone the treatment will decrease the inflammatory reaction enough to decrease length of stay and treatment and increase patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* signs/symptoms of cellulitis

Exclusion Criteria:

* steroid use in last 2 weeks
* hx of adrenal insufficiency
* suspicion for dvt or abcess
* systemic signs of sepsis
* ICU admission

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01-15 (Actual); Primary Completion 2010-08-31 (Actual); Study Completion 2010-08-31 (Actual)

PRIMARY OUTCOMES:
Time to cellulitis resolving | 48 hours after initiation of treatment

SECONDARY OUTCOMES:
Length of stay | after treatment completed

CONTACTS AND LOCATIONS:
Overall Officials: Scott Goldstein, DO, Principal Investigator — Penn State